CLINICAL TRIAL: NCT04204382
Title: Clinical Study of the Effects of Compound Kushen Injection on Radiation-induced Oral Mucositis in Head and Neck Cancer Patients.
Brief Title: Effects of CKI for Oral Mucositis Caused by Radiotherapy for Head and Neck Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanxi Zhendong Pharmacy Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDKS-CP-180503-V1.1
Record Dates: First submitted 2019-12-12; First posted 2019-12-19 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Radiation-induced Oral Mucositis
MeSH Terms: interventions — Levofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test group (Experimental): 1. CKI was injected intravenously for 7 days, once a day, 20ml each time；
  2. Levofloxacin injection were injected intravenously for 7 days, once a day, 0.5g each time,
  Interventions: Drug: Levofloxacin Injection; Drug: Compound Kushen Injection（CKI）
- control group (Other): Levofloxacin injection were injected intravenously for 7 days, once a day, 0.5g each time.
  Interventions: Drug: Levofloxacin Injection

INTERVENTIONS:
Drug: Levofloxacin Injection — Levofloxacin Injection 0.5 g each time, once a day, intravenous drip.Treatment course is 7 days.
  Other Names: Zuoyangfushaxing Zhusheye
Drug: Compound Kushen Injection（CKI） — CKI, 20mL each time, once a day, intravenous drip. Treatment course is 7 days.
  Other Names: Yanshu injection
  Arms: test group

SUMMARY:
Oral mucositis (OM) is an acute side effect of radiotherapy for head and neck cancer (HNC). OM associated pain affects oral functions and nutrition of the patient that may result in discontinuity of treatment.The purpose of this clinical study is to evaluate the therapeutic effects of Compound Kushen Injection (CKI) on oral mucositis caused by radiotherapy of head and neck cancer.

DETAILED DESCRIPTION:
Patients with oral mucositis caused by radiotherapy for Head and Neck Cancer，will be enrolled in the trial, then seprated randomly in two group,the experimental group treated with Levofloxacin injection plus CKI; the contral group treated with Levofloxacin injection only. Clinical grade of radioactive oral mucositis，Oral pain score，Completion and duration of interruption of radiotherapy， Completion of chemotherapy during concurrent chemoradiotherapy，weight change，Food intake (liquid food, semi liquid food)，recovery time of oral mucositis will be compared before treatment, 3 days, 5 days and 7 days after treatment between the experimental group and the control group.

ELIGIBILITY:
Inclusion Criteria:

1. Patients are pathologically diagnosed as stage III or stage Ⅳ squamous cell carcinoma of head and neck cancer (including nasopharyngeal carcinoma)and are in accordance with the diagnostic criteria of radiotherapy induced mucositis/ stomatitis;
2. Patients have no prior history of radiotherapy, and grade III oropharyngeal mucositis occured after the first radiotherapy;
3. Patients have no stomatological diseases such as ulcer, edema and exudation in the oropharyngeal mucosa before radiotherapy;
4. Eastern Cooperative Oncology Group (ECOG) performance Score is 0 or 1;
5. The function of each organ is basically normal, including: hemoglobins ≥ 9g/dL, platelets ≥ 80×10^9/L, leukocytes ≥ 3×10^9/L, liver function within 3 times the upper normal limit, creatinine clearance ≥ 60mL/min;
6. Patients aged between 18 and 75 years;
7. Patients have a life expectancy of at least 6 months;
8. Patients have fully understood the study and signed the informed consent voluntarily prior to any related procedures of the study.

Exclusion Criteria:

1. Patients who have received CoKS or systemic antibiotic treatment within 2 weeks before treatment;
2. Patients who have a history of head or neck surgery (except biopsy);
3. Female patients who are pregnant or breast feeding or female of pregnancy potential with a positive pregnancy test before treatment;
4. Patients with serious or uncontrolled organic diseases or infections, such as decompensate cardiac function failure, pulmonary function failure, liver function failure, renal function failure, causing unability to tolerate radiotherapy;
5. Patients who have radiotherapy contraindications;
6. Patients who are allergic to the study medications or quinolones;
7. Patients have serious psychological or psychiatric disorders, drug abuse or alcohol dependence in the past;
8. Patients are currently participating in another clinical study or have participated in another clinical trial in the past 30 days;
9. The investigator believes that it is not appropriate to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2019-12-12 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical grade of radioactive oral mucositis | From baseline to day 7.
  Treatment efficacy measured by Chinese guideline "Clinical diagnosis and treatment guidelines for tumor"
  Significant: no leukoplakia or ulcer of the oral mucosa, mild hyperemia(grade Ⅰ), able to eat regular diet.
  Effective: moderate hyperemia of the oral mucosa, mild leukoplakia or patchy ulcerations(grade Ⅱ)，semi fluid intake, but not interfering with radiotherapy.
  Ineffective: severe hyperemia of the oral mucosa, flaked leukoplakia or ulcer (grade III or above), fluid intake，severe symptoms interfering with radiation therapy , intravascular nutrition or antibiotic treatment.
  Total effective rate = (significant + effective) / total cases × 100%.

SECONDARY OUTCOMES:
Oral pain score | From baseline to day 7.
  Oral pain are evaluated with Visual Analogue Score (VAS): 0 equal no pain and 10 equal worst imaginable pain.
Completion of radiotherapy during concurrent radiotherapy | From baseline to day 7.
  Compare the proportion of patients completing radiotherapy between the two groups.
Duration of interruption of radiotherapy | From baseline to day 7.
  Compare the days of interruption period of radiotherapy between the two groups.
Completion of chemotherapy during concurrent chemoradiotherapy | From baseline to day 7.
  Compare the proportion of patients whom complete chemotherapy between the two groups.
Weight change | From baseline to day 7.
  Compare the reduction in mean weight during radiotherapy between the two groups.
Food intake (liquid food, semi liquid food) | From baseline to day 7.
  Compare intake ability of food (liquid food, semi liquid food) between the two groups.
  Effective:dietary has improved (for example, changing from liquid food to semi liquid food, from semi liquid food to soft food, or from soft food to regular diet) Ineffective: the patients can not eat, or need tube feedings, or parenteral nutrition.
Recovery time of oral mucositis | From baseline to day 7.
  Recovery time，defined as the days needs for the clinical grade of oral mucositis to fall to grade II.

CONTACTS AND LOCATIONS:
Overall Officials: Xin-xin Zhang, Principal Investigator — Chinese PLA General Hospital
Locations (12):
- China (12):
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Sun Yat-Sen Memorial Hospital Sun Yat-Sen University, Guangzhou, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong
  - Henan Anyang Tumor Hospital, Anyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - Zhenzhou Central Hospital, Zhenzhou, Henan
  - Henan Cancer Hospital, Zhenzhou, Henan
  - Affiliated Hospital of Jiangsu University, Nanjing, Jiangsu
  - Liaoning Cancer Hospital & Institue, Shenyang, Liaoning
  - Haici Medical Group, Qingdao, Shandong
  - Weihai Municipal Hospital, Weihai, Shandong
  - Second hospital of Shanxi Medical University, Taiyuan, Shanxi

IPD SHARING:
Plan to Share IPD: No